CLINICAL TRIAL: NCT04754074
Title: Diet, Food, Exercise and Nutrition During Social Distancing
Acronym: DFEND
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Jamie Baum, Associate Professor, University of Arkansas, Fayetteville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DFEND3
Record Dates: First submitted 2021-02-03; First posted 2021-02-15 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Healthy Lifestyle; Sleep; Mood; Healthy Eating
Keywords: Behavior; Nutrition; Physical activity; Diet; Exercise; Social Distancing
MeSH Terms: conditions — Behavior; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Behavioral Education and personalized coaching (Experimental)
  Interventions: Behavioral: Education; Behavioral: Personalized coaching; Behavioral: Weekly behavior modification challenges

INTERVENTIONS:
Behavioral: Education — Weekly education related to behavior change
Behavioral: Personalized coaching — Weekly calls with personalized coaches in behavior modification, nutrition, and physical activity/exercise.
Behavioral: Weekly behavior modification challenges — Weekly challenges to address behavior change

SUMMARY:
Our long-term goal is to contribute to the development of evidence-based nutritional and physical activity recommendations for the prevention and management of overweight and obesity and related chronic diseases.

The overall objective for this study is to determine if a 20-week educational program, project DFEND, related to behavior change and health will improve nutrition and physical activity outcomes as well as indicators of wellbeing.

Our central hypothesis is that regular attendance of weekly lectures, weekly meetings with personalized coaches, and weekly health challenges via virtual platforms (e.g. Zoom, Facebook, YouTube) will improve health outcomes related to nutrition and physical activity.

Our rationale for these studies is that the results of this research will enhance the potential to develop evidence-based nutritional and physical activity behavioral recommendations to treat and/or prevent development of overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Resides in Arkansas
* All ethnicities
* Female and male

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-12 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Behavior change | 20 weeks
  Participants identify one behavior they want to change and work toward achieving that goal. This will be measured by recording goals and checking in weekly to record progress. We will use a 5-point likert scale to assess how well the participant perceives they are meeting their goal. Behavior change will be assessed qualitatively, relying on the participant to report success or failures to study personnel.

SECONDARY OUTCOMES:
Sleep | 20 weeks
  Improved sleep determined by Pittsburg Sleep Quality Index questionnaire, which provides a subjective measure of sleep quality and patterns in the form of a validated questionnaire. The tool examines seven areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, the use of sleep-promoting medication, and daytime dysfunction.
Mood | 20 weeks
  Improved mood determined by Profile of Mood States questionnaire which is a psychological rating scale used to assess transient, distinct moods. It measures six different dimensions of mood swings over a period of time using a five-point scale ranging from "not at all" to "extremely".
Physical Activity | 20 weeks
  Self-reported time spent participating in physical activity using the International Physical Activity Questionnaire, which is a standardized self-report questionnaire which provides and estimate of physical activity and sedentary behavior.
Dietary Intake | 20 weeks
  Self reported diet intake using 24 hour dietary recalls

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Baum, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No